CLINICAL TRIAL: NCT02841293
Title: Cost-utility Evaluation of Two Strategies of Perineal Reconstruction After Abdominoperineal Resection for Anorectal Carcinoma: Perineal Filling With Biological Meshes vs. Primary Perineal Wound Closure
Brief Title: Cost-utility of Two Strategies of Perineal Reconstruction After Abdominoperineal Resection for Anorectal Carcinoma
Acronym: GRECCAR-9
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC31/16/7940
Record Dates: First submitted 2016-07-12; First posted 2016-07-22 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Abdominoperineal Resection
Keywords: anorectal carcinoma; perineal filling; cost-utility analysis; biological meshes; primary perineal wound closure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm with biological mesh (Experimental): The intervention consists of perinal reconstruction using biological mesh (Cellis prosthesis from Meccellis Biotech, reference C1015E size 10x15cm)
  Interventions: Procedure: Biological mesh
- Arm with primary perineal wound closure (Active Comparator): The intervention consists of perinal reconstruction by primary perineal wound closure
  Interventions: Procedure: Primary perineal wound closure

INTERVENTIONS:
Procedure: Biological mesh — The intervention consists of suturing a biological mesh in the pelvic floor defect. The mesh will be sutured at each side of the coccyx or distal sacrum and directly to the residual pelvic floor muscle and fascia by using interrupted or continuous hand-sewn sutures with an appropriate amount of tension. The mesh that will be used is the Cellis prosthesis from Meccellis Biotech, reference C1015E which size is 10x15cm.
  Arms: Arm with biological mesh
Procedure: Primary perineal wound closure — The intervention consists of stitching the ischioanal and subcutaneous fat using interrupted Vicryl sutures in one or two layers similar to primary perineal closure
  Arms: Arm with primary perineal wound closure

SUMMARY:
Abdominoperineal resection performed for anorectal tumors leaves a large pelvic and perineal defect causing a high rate of morbidity of the perineal wound (40 - 60 %). Biological meshes offer possibility for a new standard of perineal wound reconstruction. Perineal filling with biological mesh is expected to increase quality of life by reducing perineal morbidity.

DETAILED DESCRIPTION:
Perineal wound problems after abdominoperineal resection (APR) in the context of cancer are frequent. These types of resection problems occur because of wound complications caused by large perineal defects. Indeed, perineal wound complications, perineal abscess, wound dehiscences, chronic fistulas and sinuses lengthen the hospital stays. Futhermore, the standardization of the surgery since the late 2000s and the extralevator technique lead a larger defect and increase i perineal complications.

Several strategies are used to decrease the complication rate. Closure by direct approximation of the pelvic muscles leads to a rate of major complication up to 57% depending on the series. Musculocutaneous flaps help to reduce this rate (16- 65%) but they generate their own morbidity, require experience and increase the costs of care. Finally, the use of biologic meshes since the beginning of 2010 seems to have improve the healing process. However, results are still variable and the only randomized study comparing direct closure and mesh closure showed no significant results at one year. Another ongoing randomized trial is comparing gluteus maximus flap to mesh closure and focusing on physical performances.

This increase in post-operative complications and their consequences causes an increase in costs. In addition, they affect the patients' quality of life and lead to a loss of productivity. From an oncological point of view, perineal scarring problems can cause a delay in the adjuvant therapeutic sequence. Few studies have highlighted the efficiency of perineal wound complications, using cost-effectiveness analyses. In order to clarify the best strategy comparing primary and mesh closure in term of cost effectiveness on perineal healing after ELAPE, we designed this randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Eastern Cooperative Oncology Group performance status score of 2 or less
* Histologically proven rectal adenocarcinoma or anal canal epidermoïd carcinoma
* Abdominoperineal resection indication after multidisciplinary team discussion:

  * for rectal adenocarcinoma: circumferential MRI margin equal or less than 1 mm from closest tumoral structure and a striated muscular layer (levator ani or external anal sphincter)
  * for epidermoid carcinoma: residual or recurrent tumour after chemoradiotherapy.
* Voluntary written informed consent
* Patients with social security insurance or equivalent social protection

Exclusion Criteria:

* T4 tumour needing a surgical extensive resection with reconstruction by a musculocutaneous flap
* Metastasis disease deemed unresectable with curative intent
* Previous pelvic radiotherapy for another disease than the rectal or anal cancer
* Immunosuppressive drugs treatment
* Uncontrolled diabetes (glycosylated hemoglobin (HbA1c) > 8 % despite adequate therapy)
* Patient under juridical protection.
* Sensitivity to porcine derived products.
* Enrolment in trial with overlapping primary endpoint.
* Pregnant women
* Breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-02-07 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Incremental Cost-Utility Ratio (ICUR) | At 12 months
  The primary endpoint in this study is based on the assessment of the incremental cost-utility ratio at 1 year, from the collective perspective between biological mesh perineal reconstructions versus. primary perineal closure in patients operated for anorectal carcinoma with proven rectal adenocarcinoma or anal canal epidermoid carcinoma.

SECONDARY OUTCOMES:
Perineal wound healing | At 1, 3, 6, 9 and 12 months
  The perineal wound healing will be assessed using the Southampton wound assessment scale (6-point scale ranging from 0=normal healing to V=deep or severe wound infection)
Pain intensity | From date of randomization until the date of study participation end of patient, assessed up to 12 months
  assessed on an 11-point Numeric Rating Scale (NRS) at baseline before surgical procedure and at least 3 times a day during hospital stay. Thereafter, patients will rate their pain intensity in a patient subject diary every day and immediately before each use of pain medication
Health related Quality of life | 1 month, 3 months, 6 months, 9 months, 12 months
  Health related quality of life will be assessed using the EuroQOL EQ-5D-5L questionnaire
Perineal complications | Daily during hospitalization and at 1, 3, 6, 9 and 12 months after surgery
  Perineal complications include:
  * Perineal wound infection defined as a swelling of the wound or surrounding tissues with purulent discharge
  * Breakdown of the perineal wound included any wound dehiscence, sinus or ulcer
  * Pelvic abscess included a fluid collection in the pelvis
  * Perineal evisceration defined by exposure of the pelvic cavity through the perineal wound
  * Perineal hernia symptomatic or not
  * Perineal sinus defined as an incomplete healing after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Etienne BUSCAIL, MD, Principal Investigator — University Hospital of Toulouse
Locations (17):
- France (17):
  - Amiens University Hospital, Amiens
  - Angers University Hospital, Angers
  - Besançon University Hospital, Besançon
  - Bordeaux University Hospital, Bordeaux
  - Caen University Hospital, Caen
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Grenoble University Hospital, Grenoble
  - Centre Oscar Lambret, Lille
  - CHRU Lille, Lille
  - Lyon University Hospital, Lyon
  - Paoli Calmettes Institut, Marseille
  - Institut de Cancérologie de Lorraine, Nancy
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - Saint-Antoine Hospital, Paris
  - Rouen University Hospital, Rouen
  - University Hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buscail E, Canivet C, Ghouti L, Kirzin S, Carrere N, Molinier L, Rosillo A, Lauwers-Cances V, Costa N; French Research Group of Rectal Cancer Surgery (GRECCAR Group). Randomised clinical trial for the cost-utility evaluation of two strategies of perineal reconstruction after abdominoperineal resection in the context of anorectal carcinoma: biological mesh repair versus primary perineal wound closure, study protocol for the GRECCAR 9 Study. BMJ Open. 2021 Apr 1;11(4):e043333. doi: 10.1136/bmjopen-2020-043333. PMID 33795299